CLINICAL TRIAL: NCT03927014
Title: Serum Thiol/Disulphide Homeostasis Level and Its Correlation With the Severity of Preeclampsia
Brief Title: Thiol/Disulphide Homeostasis and Preeclampsia
Acronym: thiols&PE
Status: Completed | Type: Observational
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH2
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Preeclampsia
Keywords: oxidative stress; mercaptan; severity
MeSH Terms: conditions — Pre-Eclampsia | interventions — Sulfhydryl Compounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preeclampsia: The diagnosis of preeclampsia, as defined by the Committee on Terminology of the American College of Obstetricians and Gynecologists (ACOG), will establish based on the presence of proteinuria (urinary excretion of 300 mg protein or higher, or at least 1+in dipstick in a 24-h urine specimen) and a blood pressure level of ≥140/90mmHg (two blood pressure measurements 6 h apart) that occurs after 20 weeks of gestation in a previously normotensive woman. Diastolic and/or systolic blood pressure up to 110/160 mm Hg will consider mild, and higher values will consider to being severe.
  Interventions: Other: thiol/disulfide levels
- Control: The control groups' samples will obtain during the routine obstetrical care examination in the third trimester of pregnancy.
  Interventions: Other: thiol/disulfide levels

INTERVENTIONS:
Other: thiol/disulfide levels — Venous blood will sample from the antecubital veins for measuring the serum concentration of thiol/disulfide levels. The serum thiol/disulfide levels will measure using commercially available reagent kits, which is produced to detect human thiol/disulfide levels (Rel Assay Diagnostics Gaziantep, Turkey). The thiol/disulfide levels measurements were performed in accordance with the company's protocol.

SUMMARY:
Objective: To evaluate serum evaluate thiol/ disulfide levels in preeclampsia and address its relationship with its severity.

Methods: This prospective study will include 50 pregnancies complicated with preeclampsia and 50 healthy pregnancies. The blood for analysis will obtain at the admission and serum thiol/ disulfide levels will measure using commercially available reagent kits. The continuous values were evaluated using Student's t-test, and categorical values were evaluated using the Chi-square test. P values < .05 were accepted as significant.

DETAILED DESCRIPTION:
This is an observational prospective cohort study will conduct at Obstetrics and Gynecology Department of Cengiz Gokcek Obstetrics and Children's Hospital between April and October 2019. One hundred women will enrol in the study in two groups. We will consecutively recruit 50 pregnancies complicated with preeclampsia, and 50 healthy pregnancies will select for the control group. All patients will give their oral and written informed consent before their inclusion in the study. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (Reference number: 2019/147). The study strictly will adhere to the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* preeclampsia
* healthy pregnancy

Exclusion Criteria:

* pregnant women with any systemic condition (such as chronic hypertension, diabetes mellitus, thyroid diseases, liver and kidney diseases)
* women with a history of drug use throughout pregnancy
* history of medication for PE treatment at the time of first admission
* patients who had fetal congenital abnormalities or genetic syndromes
* multiple gestation
* active labor

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy
Study Population: The investigators consecutively will recruit 50 subjects with preeclampsia, and 50 healthy pregnancies will select for the control group.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Thiol/ disulfide hemostasis | 1 day
  The primary endpoint in this analysis is to evaluate thiol/disulfide levels in preeclampsia and address its relationship with its severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ovayolu, MD, Principal Investigator — Cengiz Gokcek WCH
Locations (1):
- Cengiz Gokcek Women's and Child's hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ozler S, Erel O, Oztas E, Ersoy AO, Ergin M, Sucak A, Neselioglu S, Uygur D, Danisman N. Serum Thiol/Disulphide Homeostasis in Preeclampsia. Hypertens Pregnancy. 2015 Nov;34(4):474-485. doi: 10.3109/10641955.2015.1077859. Epub 2015 Nov 20. PMID 26588703
- [Background] Yuvaci HU, Akdemir N, Bostanci MS, Yazar H, Cevrioglu S, Ozden S, Unal O, Paker MK, Neselioglu S, Erel O. Evaluation of the level of thiol-disulphide homeostasis in patients with mild and severe preeclampsia. Pregnancy Hypertens. 2016 Oct;6(4):394-399. doi: 10.1016/j.preghy.2016.09.003. Epub 2016 Sep 21. No abstract available. PMID 27939489
- [Result] Korkmaz V, Kurdoglu Z, Alisik M, Cetin O, Korkmaz H, Surer H, Erel O. Impairment of thiol-disulfide homeostasis in preeclampsia. J Matern Fetal Neonatal Med. 2016 Dec;29(23):3848-53. doi: 10.3109/14767058.2016.1149561. Epub 2016 Mar 3. PMID 26828694

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03927014/Prot_SAP_001.pdf